CLINICAL TRIAL: NCT02420197
Title: Effects of Resistance Training on Pain, Function and Work Ability in Patients With Moderate to Severe Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); Kommunal Landspensjonskasse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1157
Record Dates: First submitted 2015-03-18; First posted 2015-04-17 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Neck Pain
Keywords: Exercise therapy; Resistance training; Multidisciplinary treatment
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity resistance training (Experimental): Full body, progressive strength training with Theraband® Elastic bands. Three times per week for 12 weeks - 3 weeks with supervised sessions at the clinic, and 9 weeks of home training.Three guided sessions will be offered during the home training period.
  Interventions: Behavioral: High-intensity resistance training; Behavioral: Multidisciplinary rehabilitation program
- General physical activity (Active Comparator): 12 weeks of general physical activity - 3 weeks with supervised sessions at the clinic, and 9 weeks of individually adjusted home training. This include circle-training, low-intensity resistance exercises, endurance exercises, ball playing, body awareness, stretching, and relaxation techniques, and similar activities. Neither moderate nor high-intensity resistance exercise is included for participants in this group.Three guided sessions will be offered during the home training period.
  Interventions: Behavioral: General physical activity; Behavioral: Multidisciplinary rehabilitation program

INTERVENTIONS:
Behavioral: High-intensity resistance training
  Arms: High-intensity resistance training
Behavioral: General physical activity
  Arms: General physical activity
Behavioral: Multidisciplinary rehabilitation program

SUMMARY:
The purpose of this study is to investigate if high-intensity resistance training can induce additional beneficial effects, for patients with moderate to severe long term pain in the neck, when added to a multidisciplinary treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the multidisciplinary clinic for treatment of pain in the neck
* Long term (≥ 3months) or recurrent (≥ 2 periods of ≥ 4 weeks the past year) non-specific neck pain,
* Pain intensity ≥ 4 on numerical rating scale (0-10)

Exclusion Criteria:

* Severe somatic condition (unstable injury, malignity, infectious disease, active rheumatic disease, severe osteoporosis)
* Psychiatric condition/disease that severely impairs group functioning
* Insufficient comprehension of Norwegian language to participate in group sessions and fill out questionnaires
* Awaiting surgery of neck
* Alcohol or drug abuse
* Ongoing compensation case or applying for disability benefits due to pain in the neck
* Engaged in high-intensity resistance training on a regular basis the last 6 months
* Contra-indications for high-intensity resistance training (i.e. shoulder complications)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Neck-related disability as assessed by the neck disability index | 12 weeks
  Neck disability index

SECONDARY OUTCOMES:
Pain assessed by the Numerical Pain Rating Scale | 3 and 12 weeks + 6 and 12 months
Fear avoidance beliefs assessed by Fear Avoidance Beliefs Questionnaire | 3 and 12 weeks + 6 and 12 months
Patient's' perceived effect of the treatment assessed by the Patient specific functioning scale | 3 and 12 weeks + 6 and 12 months
Anxiety and depression assessed by Hopkins symptom checklist | 3 and 12 weeks + 6 and 12 months
Quality of life assessed by EQ-5D-5L | 3 and 12 weeks + 6 and 12 months
Work ability assessed by Work ability index | 3 and 12 weeks + 6 and 12 months
Use of analgesics assessed by a questionnaire from the HUNT study | 3 and 12 weeks + 6 and 12 months
Physical activity level assessed by a questionnaire from the HUNT study | 3 and 12 weeks + 6 and 12 months
Strength in the neck measured using a handheld dynamometer | 3 and 12 weeks + 6 and 12 months
Pressure pain threshold of the tibialis anterior muscle measured using an algometer | 3 and 12 weeks + 6 and 12 months
Grip strength measured using a handheld dynamometer | 3 and 12 weeks + 6 and 12 months
Patient's' perceived effect of the treatment assessed by the Global rating of change scale | 3 and 12 weeks + 6 and 12 months
Neck-related disability as assessed by the neck disability index | 3 weeks + 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marius S Fimland, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs University Hospital - Department of Physical Medicine and Rehabilitation, Trondheim, Norway

REFERENCES:
- [Result] Iversen VM, Vasseljen O, Mork PJ, Fimland MS. Resistance training vs general physical exercise in multidisciplinary rehabilitation of chronic neck pain: A randomized controlled trial. J Rehabil Med. 2018 Aug 22;50(8):743-750. doi: 10.2340/16501977-2370. PMID 30132009